CLINICAL TRIAL: NCT05827822
Title: Effectiveness of a WeChat-based Alcohol Consumption Intervention Mini-program ("Sober Time ACT") Among Hazardous and Problematic Drinkers in China
Brief Title: Effectiveness of a WeChat-based Alcohol Consumption Intervention Mini-program ("Sober Time ACT") in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: JDu-011
Record Dates: First submitted 2023-03-26; First posted 2023-04-25 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-03

CONDITIONS: Alcohol Use Disorder; Alcohol Abuse
Keywords: hazardous drinking; alcohol use disorders, AUDs; WeChat-based digital intervention; randomized controlled trial; mixed methods approach
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Punch-in Intervention Group (Experimental): 4 weeks of alcohol-related daily tracking + brief assessment and intervention
  Interventions: Device: Sober Time ACT
- Control Group (No Intervention): waiting list group

INTERVENTIONS:
Device: Sober Time ACT — Mental health assessment (regular assessment and reporting feedback), daily clock-in (reporting alcohol use and providing encouragement and reinforcement), mental knowledge base (Tips for the Day based on cognitive behavioral techniques, popular alcohol withdrawal courses, alcohol health education manuals) and self-assistance tools (mindfulness meditation training and emergency help buttons)
  Arms: Punch-in Intervention Group

SUMMARY:
The purpose of this study is to explore whether "Sober Time ACT", a digital intervention tool for alcohol use developed based on wechat mini program, is effective in improving risky alcohol use among Chinese local drinkers.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18
* The total score in line with the AUDIT scale ≧8
* Provide at least one backup contact information
* Non-illiterate, able to use smart phones without barriers
* Wechat version support small program function (6.5.3 and above)
* Understand the nature of this study and sign the informed consent

Exclusion Criteria:

* Other interventions and treatments to reduce alcohol use were given during the trial
* Severe primary or secondary cognitive dysfunction, unable to complete the screening scale and baseline questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Average number of risky drinking days per month | one month
  standard drinks

SECONDARY OUTCOMES:
Average weekly alcohol consumption | one month
  standard drinks
craving level | two weeks
  Pennsylvania Alcohol Craving Scale (PACS) is a single factor, multidimensional scale, Chinese version of the reliability and validity has been verified. The five items assessed frequency, intensity, duration, ability to cope with drinking and average craving on a scale of 0 to 6 points, with higher scores indicating higher craving levels.
Alcohol, Smoking, and Substance Use Involvement Screening Test (ASSIST) score | three months
  ASSIST(alcohol) was developed by the World Health Organization, based on existing screening tools, to assess risk levels for psychoactive substance use, the Chinese version has been validated for reliability and validity. There are 7 entries in the ASSIST alcohol section, and question 1 does not count towards the total score; Questions 2-5 0= never, 2= once or twice, 3= once a month, 4= once a week, 6= almost every day; Questions 6- 7,0 = never, 3= Yes but three months ago, 6= Yes in the past three months. Scores for questions 2-7 were added together to obtain an overall score for alcohol use, with 0-10 being low risk, 11-26 moderate risk, and 27+ high risk, with tertiary risk corresponding to no treatment, brief intervention, and referral to a specialist for evaluation and treatment.
willingness and confidence to abstain | one month
  The 4-item Assessment Scale of awareness, readiness and confidence in the importance of behavioral change in psychoactive substance use in the Intervention manual is scored from 0 to 10. The higher the score, the higher the degree.
stages of motivation for abstinence change | one month
  Developed by Dong Wang (2013) based on Prochaska and DiClemente's cross-theoretical model of behavioral change, It includes three dimensions: the precontemplation stage (P), the contemplation stage (C) and the action stage (A). There are 4 questions in each dimension. 1-5 points are scored. 1= strongly disagree, 2= disagree, 3= not sure, 4= agree, 5= strongly agree.
Depression, PHQ-9 | one month
  Kroenke and Spitzer (2002) revised depression screening Scale Patient Health Questionnaire, PHQ-9 based on DSM-IV diagnostic criteria, and the reliability and validity of the Chinese version have been verified (Xiaoyan Sun, Yixue Li, Canqing Yu, Liming Li, 2017). There are 9 entries, 0 to 3 on a four-point scale, 0= never at all, 1= days, 2= less than half of days, 3= almost every day. Total score 0-4 for clinically insignificant depression, 5-9 for mild depression, 10-14 for moderate depression, and 15+ for major depression.
Anxiety, GAD-7 | one month
  Generalized Anxiety Disorder, GAD-7's reliability and validity of the Chinese version of the module used to screen for generalized anxiety disorder in the Patient Health Questionnaire (PHQ) developed by Spitzer et al. (2006) (Wang Yu, Chen Ran, Zhang LAN, 2018). There are 7 entries, 0 to 3 on a four-point scale, 0= never at all, 1= days, 2= less than half of days, 3= almost every day. Total score 0-4 for clinically insignificant anxiety, 5-9 for mild anxiety, 10-14 for moderate anxiety, and 15+ for severe anxiety.
Sleep status, ISI | one month
  Insomnia Severity Index, ISI was compiled by Morin et al. (2001), the Chinese version of ISI-C has been tested to have good reliability and validity, and is suitable for the evaluation of insomnia in clinical patients in China (Bai Chunjie et al., 2018), with a total of 7 items, scoring 0-4 and 5 points. Total scores were 0-7 for nonclinically significant insomnia, 8-14 for subclinical insomnia, 15-21 for moderate clinical insomnia, and 22-28 for severe clinical insomnia.
Stress perception, PSS-10 | one month
  Perceived Stress Scale, PSS-10 is the most widely used self-assessment tool for stress feeling has high reliability and validity for the version of 10 items, 0-4 points score, 0= never, 1= rarely, 2= sometimes, 3= more, 4= very common, questions 4, 5, 7, 8 score in reverse, the higher the score indicates the higher the level of perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wu C, Yang P, Tang Y, Chen T, Li S, Huang S, Du J. Effectiveness of the WeChat-based mini-program ("Sober Time ACT") on individuals with hazardous drinking in China: a randomized controlled trial. BMC Med. 2025 Jul 1;23(1):385. doi: 10.1186/s12916-025-04217-5. PMID 40598563